CLINICAL TRIAL: NCT04685018
Title: The Neurocircuitry of Relief During Avoidance Learning in Patients With Obsessive-compulsive Disorder
Acronym: AvoidOCD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Bram Vervliet, Principal Investigator Prof. Dr. Bram Vervliet, KU Leuven
Other Study IDs: bram vervliet
Record Dates: First submitted 2020-12-14; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Avoidance behavior; Reward; Conditioning; Extinction; Anxiety Disorders; OCD; fMRI
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HC: Mentally and medically healthy adults between 18 and 60 years, free from any current or previous medical or psychiatric condition.
  Interventions: Device: fMRI acquisition
- OCD: Adults between 18 and 60 years, with a diagnosis of Obsessive-Compulsive Disorder and medication-free or with stable medication regimen for at least 3 weeks prior to the study.
  Interventions: Device: fMRI acquisition

INTERVENTIONS:
Device: fMRI acquisition — Participants from the two groups will perform an avoidance-relief task inside an MRI scanner
  Other Names: Behavioral task

SUMMARY:
To investigate the neuro-mechanisms underpinning persistent avoidance in OCD patients

DETAILED DESCRIPTION:
Many compulsions displayed by obsessive-compulsive disorder (OCD) patients serve to protect against perceived threat and can, therefore, be conceptualized as 'avoidance responses'. Exposure treatment with response prevention (ET+RP) is aimed at exposing patients to their obsessive thoughts and perceived threats while preventing engagement in compulsive avoidant responses. This induces extinction of threat perception and fearful arousal and hence reduces the motivation to avoid. While successful in many patients, however, as much as 40% dropout during treatment or display persistent avoidance after ET+RP. There is a clear need for treatment improvement for these often highly disabled patients.

Improving ET+RP outcomes requires a deeper understanding of the mechanisms that drive excessive and persistent avoidance in OCD patients. Psychological theories ascribe an important role to the relief that follows avoidance when the anticipated threat is successfully averted. This positive feeling arguably functions as a reward to reinforce the foregoing avoidance actions. Indeed, fMRI studies have found that the neurocircuitry of relief overlaps with that of reward, including the ventral tegmental area, ventral striatum and orbitofrontal cortex. Here, the authors will test the hypothesis that excessive-persistent avoidance is linked to exaggerated activation of the relief circuitry in OCD patients. For that purpose, we will acquire functional brain images of OCD patients in an MRI scanner and compare to healthy participants, while they participate in a computer task that is designed to model avoidance learning and relief.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers 18-60 years old;
* Participants are motivated and give written informed consent;
* Adequate demand of Dutch language;
* Subjects have never participated in a fear conditioning task;
* Diagnosis of OCD (for OCD group only);
* Contraindications for the MRI exam.

Exclusion Criteria:

* Current neurological (e.g. Epilepsia), respiratory, cardiovascular, metabolic, gastrointestinal, endocrine (especially diabetes), renal or urinary diseases, psychiatric disorder or other relevant medical histories (except for OCD in the OCD group);
* Being pregnant or lactating;
* Alcohol intake greater than 14 alcoholic units per week (one alcoholic unit = 10 gr ethanol);
* History of cannabis use or any other drug of abuse during the 3 months prior to the study;
* The medical doctor has asked to the participant to stay away from stressful situations;
* Electronic implants (e.g., pacemaker);
* Pain or other condition of the hand or the wrist.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy group: Mentally and medically healthy adults between 18 and 60 years, free from any current or previous medical or psychiatric condition.
  OCD group: Same as the healthy group, except for the diagnosis of OCD and medication-free or with a stable medication regimen for at least 3 weeks prior to the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2022-01-10 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Avoidance responses during the avoidance-relief task | 1 hour for avoidance task
  Avoidance responses during avoidance learning and test will be recorded in terms of button press and Reaction times
Relief during the omissions of the US | 1 hour to perform the avoidance task
  Relief will be measured as:
  Brain data during fMRI: whole-brain activations, as well as activations in specific regions of interest (ROI: VTA, NAcc, OFC) at the moment of the omissions of the electrical stimulation (US) during both the avoidance learning and the extinction learning phase of the avoidance-relief task;
  Individual ratings: relief pleasantness ratings measured on a Likert scale from 0 (neutral) to 3 (very pleasant) after each omission of the electrical stimulation (US) during both the avoidance learning and the extinction learning phase of the avoidance-relief task;
  Physiological data: skin conductance responses (SCR) at the moment of the omissions of the electrical stimulation (US) during both the avoidance learning and the extinction learning phase of the avoidance-relief task.

SECONDARY OUTCOMES:
Tolerance to stress | 1 hour to perform the avoidance task
  The individual level of tolerance to distress will be measured via the self-administration of the Distress Tolerance Scale
Therapeutic outcome in OCD | 1 hour to perform the avoidance task
  The therapeutic outcome in OCD individuals will be evaluated by using the Y-BOCS (self-administered) questionnaire
Resting-state connectivity | 1 hour to perform the avoidance task
  The strength of connectivity between NAcc, VTA, and OFC, will be measured during the resting state MRI acquisition

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatry | UZ Leuven campus Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Result] Vervliet B, Lange I, Milad MR. Temporal dynamics of relief in avoidance conditioning and fear extinction: Experimental validation and clinical relevance. Behav Res Ther. 2017 Sep;96:66-78. doi: 10.1016/j.brat.2017.04.011. Epub 2017 Apr 23. PMID 28457484
- [Result] Milad MR, Furtak SC, Greenberg JL, Keshaviah A, Im JJ, Falkenstein MJ, Jenike M, Rauch SL, Wilhelm S. Deficits in conditioned fear extinction in obsessive-compulsive disorder and neurobiological changes in the fear circuit. JAMA Psychiatry. 2013 Jun;70(6):608-18; quiz 554. doi: 10.1001/jamapsychiatry.2013.914. PMID 23740049
- [Result] Leknes S, Lee M, Berna C, Andersson J, Tracey I. Relief as a reward: hedonic and neural responses to safety from pain. PLoS One. 2011 Apr 7;6(4):e17870. doi: 10.1371/journal.pone.0017870. PMID 21490964
- [Result] Gillan CM, Morein-Zamir S, Urcelay GP, Sule A, Voon V, Apergis-Schoute AM, Fineberg NA, Sahakian BJ, Robbins TW. Enhanced avoidance habits in obsessive-compulsive disorder. Biol Psychiatry. 2014 Apr 15;75(8):631-8. doi: 10.1016/j.biopsych.2013.02.002. Epub 2013 Mar 16. PMID 23510580